CLINICAL TRIAL: NCT00016978
Title: A Phase II Study of Oxaliplatin (OXAL), 5-Fluorouracil (5-FU), and Leucovorin (CF) in Patients With Metastatic Colorectal Carcinoma Previously Treated With Irinotecan (CPT-11)
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic Colorectal Cancer Previously Treated With Irinotecan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01859; NCCTG-N9946; CDR0000068638 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-06-06; First posted 2004-03-11 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2007-08

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

ARMS (1):
- Arm I (Experimental): Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and leucovorin calcium and fluorouracil IV on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a confirmed complete response for 2 consecutive courses may discontinue study treatment at the investigators discretion. Quality of life is assessed at baseline, approximately every 6-8 weeks during treatment, and then after the last course of treatment.
  Interventions: Drug: FOLFOX regimen; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
Phase II trial to study the effectiveness of combining oxaliplatin, fluorouracil and leucovorin in treating patients who have metastatic colorectal cancer that has been previously treated with irinotecan. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the tumor response rate in patients treated with oxaliplatin, fluorouracil, and leucovorin calcium for metastatic colorectal cancer previously treated with irinotecan.

II. Determine the time to tumor progression, time to treatment failure, and overall survival of patients treated with this regimen.

III. Determine the toxicity of this regimen in this patient population. IV. Assess the quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and leucovorin calcium and fluorouracil IV on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a confirmed complete response for 2 consecutive courses may discontinue study treatment at the investigators discretion. Quality of life is assessed at baseline, approximately every 6-8 weeks during treatment, and then after the last course of treatment. Patients are followed every 3 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic colorectal adenocarcinoma incurable by surgery or not amenable to radiotherapy with curative intent
* Progressive disease no more than 3 months after completion of a prior weekly irinotecan, fluorouracil, and leucovorin calcium chemotherapy regimen
* At least 1 measurable lesion At least 20 mm in at least one dimension
* No known CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0-2
* Life expectancy: At least 12 weeks
* Absolute neutrophil count greater than 2,000/mm3
* Platelet count at least 100,000/mm3
* Bilirubin no greater than 0.5 mg/dL above upper limit of normal (ULN)
* AST no greater than 5 times ULN
* Creatinine no greater than 1.5 times ULN OR creatinine clearance greater than 60 mL/min
* No unstable angina No symptomatic congestive heart failure
* No serious uncontrolled cardiac arrhythmia
* No active or uncontrolled infection
* No evidence of other serious illness
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or noninvasive carcinomas
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No concurrent sargramostim (GM-CSF)
* At least 4 weeks since prior chemotherapy
* No more than 1 prior chemotherapy regimen for advanced colorectal cancer
* Prior adjuvant chemotherapy allowed
* No prior radiotherapy to more than 25% of bone marrow
* At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-04; Primary Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry C. Pitot, MD, Study Chair — Mayo Clinic
Locations (24):
- United States (23):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - Oncology Associates of Cedar Rapids, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada